CLINICAL TRIAL: NCT06433765
Title: BRIUMVI® Pregnancy Registry: A Prospective Study of Pregnancy and Infant Outcomes in Patients Treated With BRIUMVI®
Brief Title: A Study Evaluating the Effect of BRIUMVI® (Ublituximab) on Pregnancy and Infant Outcomes in Participants With Multiple Sclerosis (MS)
Status: Recruiting | Type: Observational
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TG1101-RMS403
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- BRIUMVI® Exposed Cohort: Pregnant participants with MS who are exposed to any dose of BRIUMVI® at any time during pregnancy (from conception to pregnancy outcome) or before pregnancy (within 6 months of the date of conception [DOC]).
  Interventions: Other: No intervention
- BRIUMVI® Unexposed Cohort: Pregnant participants with MS who are not exposed to any dose of BRIUMVI® or other anti-CD20 monoclonal antibodies at any time during pregnancy but may be exposed to other products for the treatment of MS.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The primary objective of the study is to compare the prevalence rate of major congenital malformations (MCM) between 2 cohorts of pregnant participants with MS who are exposed to BRIUMVI® and who are unexposed to BRIUMVI®.

ELIGIBILITY:
Inclusion Criteria:

1. For exposed cohort: Participant exposed to at least 1 dose of BRIUMVI®.
2. For unexposed cohort: Participants not exposed to BRIUMVI® at any time during the pregnancy.
3. Diagnosis of MS.
4. Currently or recently (within 1 year of pregnancy outcome) pregnant.
5. Authorization from healthcare provider to provide data to registry.

Exclusion Criteria:

1. Prior to enrollment, participant has exposure to anti-CD20 monoclonal antibodies at any time during pregnancy.
2. Occurrence of pregnancy outcome prior to first contact with the virtual research coordination center (VRCC) (retrospectively enrolled).
3. Exposure to known teratogens and/or investigational medications during pregnancy.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The study population will include pregnant participants with MS who are either exposed or not exposed to BRIUMVI®.
Sampling Method: Probability Sample
Enrollment: 728 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2035-03-31 (Estimated); Study Completion 2035-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Major Congenital Malformations (MCMs) | Up to 52 weeks post-delivery

CONTACTS AND LOCATIONS:
Locations (1):
- BRIUMVI® Pregnancy Registry Virtual Research Coordination Center, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No